CLINICAL TRIAL: NCT03580070
Title: Automated Multiparameter in Situ Study Comparing the Microenvironment of Head and Neck Cancers Among West Indies and Metropolitan Populations: Screening for Predictive Markers of Overall Survival and Immunotherapy Responses.
Brief Title: Changes in the Microenvironment of HPV-induced Head and Neck Cancers in West Indies and Metropolitan Population
Acronym: MituHPV
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: European Georges Pompidou Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 17/E/13
Record Dates: First submitted 2018-06-11; First posted 2018-07-09 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Immunotherapy
Keywords: Head cancers; Neck squamous cells carcinoma; HPV; Immunotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Immunotherapy — Patients with primitive head and neck squamous cells carcinoma diagnosed on surgical resection or biopsic sample, between 2008 and 2015. They were included when expressing p16 as assessed by immunochemistry and positive HPV DNA by in situ hybridation or positive HPV PCR

SUMMARY:
Retrospective observational comparative and multicentric study of the microenvironment of HPV-induced head and neck cancers, with comparison between West Indies and Metropolitan populations, and therapeutic implications. This assessment is carried out by in situ multiparametric study with multiple immunofluorescence staining for cluster of differentiation 3, cluster of differentiation 4, cluster of differentiation 8, PROGRAMMED DEATH-1, PROGRAMMED DEATH-L1, PROGRAMMED DEATH-L2, cytokeratin and cluster of differentiation 68 and automated reading. HPV genotypes will be characterized. Learning these techniques will allow me to promote them in West Indies on my way back, and they may be applicable to other HPV-induced cancers.

DETAILED DESCRIPTION:
Global annual incidence of head and neck (HN) cancers is high. It is even a greater concern in West Indies compared to other American countries. Most represented histological type is squamous carcinoma and several risk factors are involved , including tobacco exposure. Moreover, it is now clear that Human Papillomavirus (HPV) is a causal factor in the development of HNSCCs : as many as 5 to 10% of tumors are induced by HPV in the world, and it is responsible of 25,9% of HN tumors. HPV 16 is the most involved (87%). However, HPV epidemiology is different in West Indies with the implication of various genotypes. Detection of HPV infection can be achieved through several methods such as polymerase chain reaction (PCR) or RNAscope, which is a new reliable precise technique which reflects the transcriptional activity of the virus. The differences between the genotype of HPV involved within both populations need to be consider to better identify therapeutic targets.Studying the microenvironment may allow a better understanding of anti-tumoral immunity and may help patient selection in order to achieved better responses to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Primitive head and neck squamous cells carcinoma diagnosed on surgical resection or biopsic sample, between 2008 and 2015 in metropolitan and Antillean populations. For metropolitan they were included when expressing p16 as assessed by immunochemistry and positive HPV DNA by in situ hybridation or positive HPV PCR. For Antillean population they were included when expressing p16 as assessed by immunochemistry with regards of genotype as assessed by in situ hybridation or by PCR (to be completed).

Exclusion Criteria:

* Secondary tumors,
* Tumor recurrence in a patient for whom we have already tumor tissue, nasopharyngeal tumors, p16 expression by immunochemistry with negative PCR testing for HPV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with primitive head and neck squamous cells carcinoma diagnosed on surgical resection or biopsic sample, between 2008 and 2015 in metropolitan and Antillean populations
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Description of tumoral microenvironment with multiparametric study by immunofluorescence comparing West Indies population and metropolitan population and the stratification of patients regarding RNAscope staining intensity and HPV genotype. | 12 months
  Automated reading of results by software Inform (Perkin©).

SECONDARY OUTCOMES:
The secondary outcome measures are: - interpretation of RNAscope results and comparison between West Indies and Metropolitan population, - evaluation of RNAscope staining intensity to define subgroups | 12 months
  Automated reading of results by software Inform (Perkin©).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MOLINIE, Pr, Principal Investigator — CHU Martinique
Locations (2):
- Hôpital Européen Georges Pompidou, Paris, France
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No